CLINICAL TRIAL: NCT00177723
Title: Towards Reducing Resistance and Hematological Toxicity of Linezolid
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: Monash University (Other)
Other Study IDs: IRB# 0501019
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2008-12-17 (Estimated); Status verified 2008-12

CONDITIONS: Infection; Adverse Effects
Keywords: receiving antibiotic Linezolid clinically
MeSH Terms: conditions — Infections

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
The study will evaluate and improve the performance of pharmaco-statistical models previously developed in the compassionate use program in patients being treated with linezolid under clinical usage conditions. This study will also develop a sensitive and specific tool that may be used to predict patients at risk of hematological toxicity, based on factors including linezolid concentration and duration of therapy and use these models to better understand the determinants of toxicity with linezolid and define better strategies to manage toxicity or reduce its occurrence.

DETAILED DESCRIPTION:
Epidemiologic information to be collected

At baseline (upon signing informed consent), the following information will be collected: Demographic data - age, sex, height, weight, state of birth, previous pathology reports associated with the bacteria the subject has contracted, laboratory results, current medication use, and any other prior medical problems/history. The following outcome measures will be assessed: (a) time to resolution of fever, (b) time to normalization of white blood cell count, (c) time to microbiologic eradication of infection, (d) mortality at 28 days following onset of infection.

Blood work to be collected

Hematological parameters:

Patients included in this study will be required to have blood samples taken to determine their platelet count and hemoglobin at baseline (prior to the first dose of linezolid), weekly whilst receiving linezolid and at end of linezolid treatment. Monitoring of hematological parameters is recommended as part of the standard of care for patients being treated with linezolid for greater than 2 weeks. This information will be collected from the participant's medical record and become part of the research record.

Pharmacokinetic samples:

On doses 4 or 5 of Linezolid administration blood samples will be obtained from the patient's vein prior to the first dose of the day of intravenous (IV) or oral Linezolid. Subsequent samples of blood will be obtained over an eight hour period following dose administration (2 hours, 4 hours and 8 hours after dose administration). About 5 ml or one teaspoon will be obtained by the bedside nurse for each blood sample for a total of 20 ml or 4 teaspoonfuls. The GCRC staff will travel to the patient's hospital unit and obtain the blood samples when necessary. If the patient is an outpatient, the patient will be asked to come to the GCRC to have the blood samples withdrawn.

If the samples are not obtained prior to the first dose of medicine on days 2 or 3 of dose administration, blood can be obtained from the patient's vein around two separate doses on day 2 and 3 and day 3 and 4. Blood will be obtained from the patient's vein prior to taking the next dose of IV or oral Linezolid and two hours after the medicine has been administered. About 10 ml or two teaspoonfuls will be obtained by the bedside nurse for each blood sample for a total of 20 ml or 4 teaspoonfuls.

If the patient develops a decrease in hematologic parameters (defined as Hb < 10 g/dL, WBC < 2.5, ANC <1.5 or platelets <100), blood will be collected from the patient's vein immediately before a linezolid dose and two hours after the medicine has been administered. At these levels, the clinicians caring for the patient will be advised that the frequency of hematologic monitoring should increase to three times weekly. If the following hematologic parameters occur, the clinician will be advised by the investigators to consider utilizing an alternative antibiotic: Hb <8 mg/dL, WBC <1.5, ANC <1.0, platelets <50. It is acknowledged that the investigators are not responsible for the care of the patient and that many factors may influence the clinician's decision to continue or to switch linezolid therapy. The management decisions will be made by the patient's clinical team and NOT the investigators.

The blood samples will be processed and stored in a - 80° C freezer in a secured laboratory under the supervision of the principal investigator. These samples will then be used to determine the amount of Linezolid that reached the participant's blood following dose administration.

All samples will be analyzed to obtain the amount of Linezolid found in the blood. No genetic testing will be performed on any of the samples being obtained. The biologic samples (blood) will be under the control of the principal investigator of this research project. To protect confidentiality, all personal identifiers (i.e., name, social security number, and birth date) will be removed (de-identified) and replaced with a specific code number. The information linking these code numbers to the corresponding subjects' identities will be kept in a separate, secure location. The investigators on this study will keep the samples indefinitely. Part of the biologic samples will be sent to Dr. Craig Rayner at Monash University of Australia. All samples sent outside of the UPMC facility will be de-identified. Samples sent to Monash University will be kept in Dr. Rayner's laboratory. If a subject withdraws and provides the request in writing, samples collected and not already processed will be destroyed. All samples at UPMC will be kept in the investigator's laboratory located in Scaife Hall, Room 812, 3550 Terrace Street.

All patients will be seen at the UPMC facility while they are inpatients.

If a subject is removed from Linezolid clinically, subjects will not be required to prolong the use of Linezolid and the subject's hospitalization will not be prolonged if not clinically indicated.

ELIGIBILITY:
Inclusion Criteria:

* Males or females greater than 18 years of age.
* All patients will remain in the hospital for pharmacokinetic sampling.
* All subjects must be on the medication linezolid as part of their standard of care.

Exclusion Criteria:

* Patients with renal failure who receive peritoneal dialysis, hemodialysis or hemofiltration.
* Any contraindication to blood sampling

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2005-08; Study Completion 2007-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David L Paterson, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States